CLINICAL TRIAL: NCT07174076
Title: Prevention of Recurrence With Cordyceps Sinensis in Mycobacterium Avium Complex Pulmonary Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bin Cao (Other)
Collaborators: China-Japan Friendship Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Jiangxi Chest Hospital (Unknown); Guangzhou Chest Hospital. (Unknown); Anhui Chest Hospital (Other); Beijing Chest Hospital (Other); Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Bin Cao, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025-KY-004-1
Record Dates: First submitted 2025-07-22; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Mycobacterium Avium Complex Pulmonary Disease
Keywords: mycobacerium avium complex; recurrence; cordyceps sinesis
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cordyceps sinesis (Experimental): cordyceps sinesis capsule 4# tid for 12 months
  Interventions: Drug: cordyceps sinesis capsule
- Placebo (Placebo Comparator): placebo 4# tid for 12 months
  Interventions: Drug: cordyceps sinesis capsule placebo

INTERVENTIONS:
Drug: cordyceps sinesis capsule — cordyceps sinesis capsule 4 capsules tid po for 12 months
  Arms: Cordyceps sinesis
Drug: cordyceps sinesis capsule placebo — cordyceps sinesis capsule placebo 4 capsules tid po for 12 months
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if cordyceps sinesis capsule (Bailiing Capsule) works to prevent the recurrence of microbiologically cured mycobacterium avium complex pulmonary disease in adults. The main questions it aims to answer are:

Does cordyceps sinesis capsule (Bailiing Capsule) prevents the recurrence of mycobacterium avium complex pulmonary disease in adults? Researchers will compare cordyceps sinesis capsule (Bailiing Capsule) to a placebo (a look-alike substance that contains no drug) to see if cordyceps sinesis capsule helps to prevent the recurrence of mycobacterium avium complex pulmonary disease.

Participants will:

Take cordyceps sinesis capsule (Bailiing Capsule) or a placebo (a look-alike substance that contains no drug) for 12 months, both are administered every day.

Visit the clinic once every 3 months for checkups and tests. Take online questionnaires every month.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in the study and sign the informed consent form.
2. Age between 18 and 75 years, inclusive; gender unrestricted.
3. Confirmed diagnosis of MAC (Mycobacterium avium complex) lung disease according to either the 2020 ATS/IDSA guidelines or the Chinese Guideline for Diagnosis and Treatment of Nontuberculous Mycobacterial Disease (2020 edition). Imaging findings at baseline must show a nodular bronchiectatic pattern prior to treatment initiation.
4. Completed the recommended treatment regimen for nodular-bronchiectatic MAC lung disease (macrolide + ethambutol + rifampin, with minimum 12-month duration) per the above guidelines within 3 months prior to screening; Fully completed the anti-infective treatment phase of this study. Participants must achieve bacteriologic negativity (two consecutive negative sputum cultures with an interval ≥4 weeks) by the end of their treatment course.
5. For non-surgically sterilized women of childbearing potential:

   Must use a medically approved contraceptive method (e.g., intrauterine device, hormonal contraceptives, or condoms) during the study period and for 3 months post-last treatment dose. A negative serum/urine pregnancy test must be confirmed within 72 hours prior to enrollment.

   Must not be lactating at screening.

   For male participants with partners of childbearing potential:

   Must use effective contraception during the study and for 3 months post-last treatment dose.
6. Organ Function Requirements (Met Within 1 Week Prior to Enrollment):

i. Hemoglobin ≥60 g/L; ii. Neutrophil count ≥0.5 × 10⁹/L; iii. Platelet count ≥60 × 10⁹/L; iv. Serum total bilirubin ≤3× upper limit of normal (ULN); v. Aspartate aminotransferase (AST) ≤3× ULN; vi. Alanine aminotransferase (ALT) ≤3× ULN; vii. Serum creatinine <2× ULN or creatinine clearance ≥60 mL/min; viii. Blood urea nitrogen (BUN) ≤200 mg/L; ix. Urine protein <++ on dipstick; if trace (+), 24-hour urine protein must be <500 mg; x. Fasting glucose within normal range **or** controlled stable glycemic levels in diabetic patients; xi. Cardiac function: No myocardial infarction in the past 6 months, no unstable angina, no severe arrhythmias, and New York Heart Association (NYHA) functional class ≤II.

Exclusion Criteria:

1. Any allergy to drugs included in the treatment regimen.
2. Completed anti-MAC therapy for more than 3 months.
3. Active respiratory tract infection.
4. Presence of congenital/acquired immunodeficiency diseases, active pulmonary malignancies (primary or metastatic), or any malignant tumors requiring chemotherapy/radiotherapy during screening or the study period.
5. History of solid organ transplantation.
6. Currently undergoing dialysis.
7. Radiographic pneumonia requiring steroid/immunoglobulin pulse therapy, clinically evident active interstitial lung disease, uncontrolled massive pleural effusion/pericardial effusion.
8. Unstable concomitant systemic diseases (hypertensive crisis, unstable angina, congestive heart failure, myocardial infarction within the past 6 months, severe psychiatric disorders requiring medication, severe hepatic/renal dysfunction, neurodegenerative diseases such as Alzheimer's disease).
9. Poor gastrointestinal function or malabsorption syndrome.
10. Receipt of other investigational drugs (excluding participation of 2025-KY-004-1) within 4 weeks prior to the first administration of study drug.
11. Participation in another interventional clinical trial simultaneously, except for observational/non-interventional trials or follow-up periods of interventional trials.
12. Any physical examination findings or clinical laboratory results that the investigator believes may interfere with study outcomes or pose increased risks of complications for the patient's management.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2028-07-24 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
bacterial recurrence of MAC-PD | from enrollment to the end of month 12

SECONDARY OUTCOMES:
occurrence of respiratory infection | from enrollment to the end of month 12

OTHER OUTCOMES:
adverse events and laboratory findings | from enrollment to the end of month 12
recurrent MAC strain subtype | from enrollment to the end of month 12

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Cui, M.D., Principal Investigator — China-Japan Friendship Hospital
Locations (6):
- China (6):
  - Anhui Chest Hospital, Hefei, Anhui
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Guangzhou Chest Hospital, Guangzhou, Guangdong
  - Jiangxi Chest Hospital, Nanchang, Jiangxi
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No